CLINICAL TRIAL: NCT05856279
Title: Immediate Effect of Two Selected Mulligan Techniques on Lumbar Sagittal Mobility in Nonspecific Low Back Pain
Brief Title: Immediate Effect of Two Selected Mulligan Techniques in Nonspecific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samaa Atef Abd Elazeez Mohamed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004356
Record Dates: First submitted 2023-04-15; First posted 2023-05-12 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Back Pain
Keywords: mulligan; lumbar; sagittal; mobility; Back; pain
MeSH Terms: conditions — Back Pain; Pain | interventions — Movement

STUDY DESIGN:
Intervention Model Description: mulligan SNAG and mulligan lion position
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded clinical randomized controlled trial (research assistant for assessment and patients will be blinded to about treatment).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mulligan SNAG (Experimental): Patients in this group will receive mulligan SNAG from sitting position and McGill stabilization exercises.The glide will be performed six repetitions for three sets for one session and McGill stabilization exercises as a home program: 7 days a week and 10 repetitions of each exercise for 2times per day and a rest interval of 2 minutes between exercises
  Interventions: Procedure: mulligan SNAG and mulligan lion position
- mulligan lion position (Experimental): Patients in this group will receive mulligan modified lumbar SNAG lion position and McGill stabilization exercises.Modified lumbar SNAGs (lion position) will be applied in a quadruped position (lion position)six repetitions for three sets for one session . McGill stabilization exercises as a home program: 7 days a week and 10 repetitions of each exercise for 2times per day and a rest interval of 2 minutes between exercises The therapist stands to one side of the patient and applies (SNAG) centrally to the spinous process of the involved segment. The medial border of the hand is hooked under the chosen segment while the other arm encircles the trunk to stabilize the upper body. The therapist maintains the glide while the patient sits back towards their heels (for flexion) .
  Interventions: Procedure: mulligan SNAG and mulligan lion position

INTERVENTIONS:
Procedure: mulligan SNAG and mulligan lion position — manual therapy techniques for lumbar spine
  Other Names: moblization with movement

SUMMARY:
To compare between immediate effect of SNAG and mulligan lion position in range of motion (ROM) , pain, functional ability and kinesiophobia on patients with nonspecific low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is a global health problem.Orthopedic Manual therapy (OMT) is most commonly recommended form of treatment of LBP and it is also frequently used in clinical practice in various countries. Mulligan introduced a new technique in manual therapy. Mulligan has a great role in the treatment of LBP.General techniques of mulligan are MWM, SNAGs and natural apophyseal glides (NAGs).

Lumber SNAG have immediate and short term on pain and function in treatment of patients with NSLBP.Mulligan has special techniques, one of them is modified lumbar SNAG (lion position) .It has short term effect in reducing pain and activity limitation. Up to investigated knowledge, No previous studies comparing immediate effect of two techniques in range of motion (ROM), pain, functional ability and kinesiophobia

ELIGIBILITY:
Inclusion Criteria:

1. 3 to 7 on VAS.
2. Back Pain duration of 6 week or more .
3. 20-40 years old .
4. Patients of both sexes will be concluded .
5. body mass index (18.5-29.9 KG/M2).

Exclusion Criteria:

1. fracture, osteoporosis, myelopathy, multiple adjacent radiculopathies, cauda equina syndrome, vertebral bone disease and bony joint instability .
2. Infective conditions of spine, autoimmune disorders, Pacemakers, malignancy .
3. History of surgery or injection at lumbar spine 1 year ago .

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
ROM | up to 2 hours after technique
  ROM by bubble inclinometer

SECONDARY OUTCOMES:
degree of Pain | one week
  Pain will be assessed by VAS.

OTHER OUTCOMES:
Functional disability | one week
  Functional disability will be assessed by the arabic version of Oswestry
Kinesiophobia | one week
  Kinesiophobia will be assessed Tampa scale -Arabic version

CONTACTS AND LOCATIONS:
Overall Officials: samaa Mohammed, Principal Investigator — physical therapist at Badr central hospital
Locations (1):
- Samaa Atef Abd El Azeez Mohammed, Beheira, Egypt